CLINICAL TRIAL: NCT04649775
Title: AirFLO2 Treatment for Hypoxia and/or Tachypnea in Patients With COVID-19
Acronym: AirFLO2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no eligible participants
Sponsor: Duke University (Other)
Collaborators: MEDEX (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105246
Record Dates: First submitted 2020-10-14; First posted 2020-12-02 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-04

CONDITIONS: Corona Virus Infection; Respiratory Rate; Hypoxia; Covid19
MeSH Terms: conditions — Coronavirus Infections; Hypoxia; COVID-19

STUDY DESIGN:
Intervention Model Description: Unblinded, randomized, controlled trial with two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Device intervention (Active Comparator): Intervention participants will receive the AirFLO2 device and training via video with reinforcement from the coordinator how to use and to self-apply it. Clinical data will be recorded before and after intervention. Questionnaires will be completed at baseline and at serial time points after intervention starts.
  Interventions: Device: AirFLO2
- Standard of Care- Control (No Intervention): Participants will receive standard of care, clinical data will be recorded. Baseline and end of study questionnaires will be performed.

INTERVENTIONS:
Device: AirFLO2 — Mask device
  Arms: Device intervention

SUMMARY:
The study is an unblinded, randomized, controlled trial for use of the AirFlO2 device for patients admitted to Duke Hospital with COVID-19 and tachypnea (RR >20 breaths/min) and/or hypoxia (Oxygen saturation <94% on room air or requiring supplemental oxygen at baseline).

DETAILED DESCRIPTION:
The aim of the study is to determine whether the use of the AirFLO2 device can improve hypoxia as measured by change between partial pressure of arterial oxygen to fraction of inspired oxygen- P:F ratio (PaO2:FiO2) and repeat P:F ratio between 1 to 6 hours after using the device.

This is an unblinded, randomized, controlled trial for use of the AirFLO2 device for patients admitted to Duke Hospital with COVID-19 and tachypnea (RR >20 breaths/min) and/or hypoxia (Oxygen saturation <94% on room air or requiring supplemental oxygen at baseline).

Groups will be analyzed by intention to treat. Per-protocol analyses will also be performed. Descriptive statistics will be reported for the overall subject population, and for the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age with confirmed COVID-19 infection
* Patient must be able to complete consent and hold mask
* Baseline room air oxygen saturation <94% or new supplemental oxygen requirement at presentation or patient on supplemental oxygen at baseline and requiring up-titration of oxygen setting
* Patient in negative pressure room
* Patient must have access to an internet-connected device

Exclusion Criteria:

* Tracheostomy
* History of pneumothorax or known bullous lung disease
* Recent cataract surgery
* Patient receiving NIV (Noninvasive Ventilation) or HFNC (High Flow Nasal Cannula)
* Patient receiving mechanical ventilation
* Delirium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Que, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AirFLO2 Device Intervention: Intervention participants will receive the AirFLO2 device and training via video with reinforcement from the coordinator how to use and to self-apply it. Clinical data will be recorded before and after intervention. Questionnaires will be completed at baseline and at serial time points after intervention starts.
  AirFLO2: Mask device
- Standard of Care - Control: Participants will receive standard of care, clinical data will be recorded. Baseline and end of study questionnaires will be performed.
Period: Overall Study
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.8) | 42.1 (9.8) | 47.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Oxygenation as Measured by P:F Ratio (PaO2:FiO2)
Description: A higher P:F ratio value indicates better oxygenation. Range 20 to 500.
Time Frame: Baseline, 24 hours, 48 hours
Population: Data not collected at 48 hours on two participants in the Standard of Care - Control arm.
Measure: Mean (Standard Deviation); unit: P:F ratio
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 6
P:F ratio
  Baseline | 250.5 (35.0) | 272.8 (44.9)
  24 hours | 275.6 (61.0) | 264.2 (48.8)
  48 hours: number analyzed (Participants) | 5 | 4
  48 hours | 253.9 (64.7) | 263.0 (100.8)

2. Secondary Outcome: Subject Dyspnea Symptoms
Description: Improved symptoms related to dyspnea as measured by the change in the Modified Medical Research Council (MMRC).. Range 0 to 4 with lower values being better.
Time Frame: baseline to end of hospitalization (discharge from hospital or death, 1 - 30 days range)
Population: Data not collected.
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Participant Cough Symptoms as Measured by the Leicester Cough Questionnaire (LCQ)
Description: The Leicester Cough Questionnaire (LCQ) questionnaire has a score range of 3-21, where a higher score indicates better quality of life.
Time Frame: baseline to up to six hours for device intervention participants; baseline to hospital discharge (up to 30 days) for all patients
Population: Data not collected for one participant in the Standard of Care - Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 5
score on a scale | 8.00 (4.74) | 5.60 (2.79)

4. Secondary Outcome: Change in Participant Respiratory Symptoms as Measured by the St George Respiratory Questionnaire (SGRC)
Description: The St George Respiratory Questionnaire (SGRC) questionnaire has a score range of 0-100, where a higher score indicates worse quality of life.
Time Frame: as for outcome 3
Population: Data not collected on one participant in the Standard of Care - Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 5
score on a scale | -25.33 (20.61) | -23.38 (24.00)

5. Secondary Outcome: Number of Participants Transferred to High Flow Nasal Cannula (HFNC), Non-invasive Ventilation (NIV), or Invasive Ventilation
Description: Reduce risk of respiratory deterioration as measured by change from baseline to end of hospitalization (discharge or patient death) to high flow nasal cannula (HFNC), non-invasive ventilation (NIV), or invasive ventilation.
Time Frame: baseline to end of hospitalization (discharge from hospital or death, 1 - 30 days range)
Measure: Count of Participants; unit: Participants
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 6
Participants
  Transfer to HFNC | 2 | 1
  Transfer to NIV | 0 | 0
  Transfer to ventilation | 0 | 0

6. Secondary Outcome: Number of Participants Transferred to the ICU
Description: Reduced intensive care unit (ICU) transfer risk occurring between baseline and end of hospitalization
Time Frame: baseline to end of hospitalization, (discharge from hospital or death, 1 - 30 days range)
Population: Data not collected at 48 hours on two participants in the Standard of Care - Control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 6
Participants
  24 hours | 0 | 0
  48 hours: number analyzed (Participants) | 5 | 4
  48 hours | 0 | 1

7. Secondary Outcome: Number of Participants Requiring Intubation
Description: Reduce risk for intubation requirement as measured by incidence of intubation occurring between baseline and end of hospitalization (discharge or death)
Time Frame: baseline to end of hospitalization (discharge from hospital or death, 1 - 30 days range)
Measure: Count of Participants; unit: Participants
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

8. Secondary Outcome: Hospitalization Length of Stay in Days
Description: Hospitalization length of stay as measured by length of hospitalization after the baseline timepoint.
Time Frame: baseline to end of hospitalization (discharge from hospital or death, 1 - 30 days range)
Measure: Mean (Full Range); unit: days
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 6
days | 6.6 [4 to 8] | 9.0 [3 to 32]

9. Secondary Outcome: Number of Participants Who Survived to Discharge
Description: Patient survival to hospital discharge as measured by the participant status at the end of the hospitalization (discharge or death)
Time Frame: baseline to end of hospitalization (discharge from hospital or death, 1 - 30 days expected range)
Measure: Count of Participants; unit: Participants
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
Number analyzed (Participants) | 5 | 6
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: Baseline to end of hospitalization, up to approximately 30 days
Arm/Group | AirFLO2 Device Intervention | Standard of Care - Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT04649775/Prot_SAP_000.pdf